CLINICAL TRIAL: NCT04677933
Title: A Phase 1b, Randomised, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Multiple Subcutaneous Doses of OLP-1002 in Patients Who Have Pain Due to Moderate to Severe Osteoarthritis in a Hip and/or Knee Joint
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Multiple Subcutaneous Doses of OLP-1002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OliPass Australia Pty Ltd (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OLP-1002-001B
Record Dates: First submitted 2020-11-17; First posted 2020-12-21 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Patients will receive 5 µg OLP-1002 BIW for 15 days (Day 1, 4, 8, 11 and 15). Mode of Administration: Subcutaneous injection
  Interventions: Drug: A: OLP-1002
- Arm B (Experimental): Patients will receive 10 µg OLP-1002 BIW for 15 days (Day 1, 4, 8, 11 and 15). Mode of Administration: Subcutaneous injection
  Interventions: Drug: B: OLP-1002
- Arm C (Experimental): Patients will receive Diluent placebo BIW for 15 days (Day 1, 4, 8, 11 and 15) Mode of Administration: Subcutaneous injection
  Interventions: Drug: C: Placebo

INTERVENTIONS:
Drug: A: OLP-1002 — 10 patients will receive 5 µg OLP-1002 twice-weekly (BIW) OLP-1002
  Other Names: OLP-1002: A
  Arms: Arm A
Drug: B: OLP-1002 — 10 patients will receive 10 µg OLP-1002 BIW OLP-1002
  Other Names: OLP-1002: B
  Arms: Arm B
Drug: C: Placebo — 10 patients will receive Placebo BIW
  Other Names: Placebo
  Arms: Arm C

SUMMARY:
This is a Phase 1b, randomised, double-blind, placebo-controlled, parallel study to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of multiple SC doses of OLP-1002 in patients who have pain due to moderate to severe osteoarthritis (OA) in a hip and/or knee joint. The study consists of:

* Screening period: up to 14 days (defined as Day -23 to -9)
* Washout period: 5 days (± 1 day) (defined as Day -8 to -4)
* Baseline period: 3 days (± 1 day) (defined as Day -3 to -1, where Day -1 is the day before dosing)
* Treatment period: 15 days (± 1 day) (defined as Day 1 to 15, where Day 1 is the day of first dosing)
* Follow-up period: 30 days (± 5 days) (defined as Day 16 to 45, assuming Day 15 is the day of the last dose)

Up to 30 patients will be enrolled in the study and will be randomised in the ratio 1:1:1 to the following arms:

* Arm A: 10 patients will receive 5 µg twice-weekly (BIW) OLP-1002
* Arm B: 10 patients will receive 10 µg BIW OLP-1002
* Arm C: 10 patients will receive Placebo BIW

DETAILED DESCRIPTION:
Study drug: OLP-1002

Proposed Dose:

1. 5 microgram twice a week (BIW) for 15 days (Day 1, 4, 8, 11 and 15)
2. 10 microgram BIW for 15 days (Day 1, 4, 8, 11 and 15)

Mode of Administration: Subcutaneous injection

The study will consist of 5 time periods:

* Screening period: up to14 days
* Washout period: 5 days (± 1 day)
* Baseline period: 3 days (± 1 day)
* Treatment period: 15 days (± 1 day)
* Follow-up period: 30 days from last dose (± 5 days)

Up to 30 patients will be enrolled in the study and will be randomised in the ratio 1:1:1 to the following arms:

* Arm A: 10 patients will receive 5 µg BIW OLP-1002
* Arm B: 10 patients will receive 10 µg BIW OLP-1002
* Arm C: 10 patients will receive Placebo BIW

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged greater than or equal to 35 years to lesser than or equal to 65 years as of the date of study enrolment;
2. Patients must be willing and able to provide written informed consent after the nature of the study has been explained and prior to the commencement of any study procedures;
3. Patients have a BMI greater than or equal to 18 and less than 40 kg/m2 at Screening;
4. Patients have pain in (a) hip or knee joint/s, every day for at least one month during the three months prior to Screening;
5. Patients have a diagnosis of moderate to severe OA of the index hip or knee: moderate to severe osteoarthritis, based on American College of Rheumatology (ACR) criteria with Kellgren Lawrence X-ray grade of at least 3 as diagnosed by the radiologist;
6. Patients with WOMAC Total Pain subscale score of ≥ 10 in the index hip or knee at Screening;
7. Patients who are willing to discontinue all non-study pain medications except for permitted rescue pain medication for the duration of the study;
8. Patients agree to maintain their usual levels of activity throughout the course of the study and until End of Study (EOS) (Day 45);
9. Patients who are willing to abstain from all other intra-articular treatments of the joint and any joint surgery while in the study and until EOS (Day 45);
10. Patients having clear injection sites, although parts of the body have tattoos;
11. Patients who are willing and able to comply with study procedures, including the recording of daily questionnaires;
12. Females must be non-pregnant and non-lactating, and must use acceptable, highly effective double contraception from screening until 90 days after the last dose of study drug. Double contraception is defined as a condom AND one other form of the following:

    1. Established hormonal contraception (for example, approved oral contraceptive pills (OCPs), long-acting implantable hormones, injectable hormones);
    2. A vaginal ring or an intrauterine device (IUD); or
    3. Documented evidence of surgical sterilisation at least 6 months prior to screening (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, or bilateral oophorectomy for women or vasectomy for men [with appropriate post-vasectomy documentation of the absence of sperm in semen] provided the male partner is a sole partner)
    4. Women not of childbearing potential must be post-menopausal for ≥12 months. Post-menopausal status will be confirmed through testing of follicle-stimulating hormone (FSH) levels ≥ 40 IU/mL at Screening for amenorrhoeic female patients. Females who are abstinent from heterosexual intercourse will also be eligible.
    5. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not considered highly effective methods of birth control. A patient's complete abstinence for the duration of the study and for 90 days after the last study treatment is acceptable.
    6. Female patients who are in a same-sex relationships are not required to use contraception.
    7. Males must be surgically sterile (greater than 30 days since vasectomy with no viable sperm), abstinent, or if engaged in sexual relations with a women of child bearing potential (WOCBP), the patient and his partner must be surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or using an acceptable, highly effective contraceptive method from Screening until 90 days after the last dose of study drug. Acceptable methods of contraception include the use of condoms and the use of an effective contraceptive for the female partner that includes: OCPs, long acting implantable hormones, injectable hormones, a vaginal ring or an IUD. Patients with same-sex partners (abstinence from penile-vaginal intercourse) are eligible when this is their preferred and usual lifestyle;
13. WOCBP must have a negative pregnancy test at Screening and Day 1 and be willing to have additional pregnancy tests as required throughout the study;
14. Males must not donate sperm for at least 90 days after the last dose of study drug.

Exclusion Criteria:

1. Any of the following:

   * QTcF greater than 450 ms confirmed by repeat ECG measurement
   * QRS duration greater than 110 ms confirmed by repeat ECG measurement
   * PR interval greater than 220 ms confirmed by repeat ECG measurement
   * Findings which would make QTc measurements difficult or QTcF data uninterpretable
   * History of additional risk factors for torsades de pointes (e.g., heart failure (class III/IV according to the New York Heart Association [NYHA]), hypokalaemia, family history of long QT syndrome)
2. Intraarticular treatment injections (including but not limited to corticosteroids, hyaluronic acid, platelet rich plasma, BOTOX®, local anaesthetics) within 3 months prior to the Screening period
3. Patients who are unable or unwilling to cease the use of all pain medications, prescription, over-the-counter and otherwise, as of the first day of the study Washout Period and until after Day 45 of the study. This includes all opioid and anti-inflammatory medications. This excludes the use of paracetamol provided that a patient is able and willing to utilise a maximum of 2 g of paracetamol per 24-hour period as of the first day of the study Washout Period and until after Day 45 of the study, unless the PI has approved an increased dose up to 4 g;
4. Use or intend to use TENS machine during the study period, i.e. from screening until after Day 45 of the study;
5. Any of the following laboratory abnormalities within 14 days of the first treatment day:

   * Platelet count less than 100,000 cells/mm3
   * Total neutrophil count less than 1,500 cells/mm3
   * Serum creatinine greater than or equal to 1.5 x ULN
   * Alanine aminotransferase (ALT) greater than 3.0 x ULN
   * Aspartate aminotransferase (AST) greater than 3.0 x ULN
   * Alkaline phosphatase greater than 2.0 x ULN
   * Bilirubin greater than 1.5 x ULN
   * Temperature greater than or equal to 38°C or any other evidence of an infection
6. History of alcohol or substance abuse or dependence during the 12 months prior to Screening

   * During the study, alcohol consumption of greater than 21 units per week for males and greater than14 units per week for females will not be allowed. One unit of alcohol equals ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits;
   * Positive urine drug screen (confirmed by repeat) or alcohol consumption (self-report) higher than the permissible limit, as mentioned above, within the preceding 3 days at Screening or Baseline shall be excluded from the study;
7. Use or intend to use medication that interacts with CYP3A4 and/or CYP2D6.
8. Has an allergy or hypersensitivity to the study drug or its components;
9. Female patients who are pregnant at Screening or are planning on becoming pregnant, or are currently breastfeeding;
10. Patients with any medical condition or comorbidities that could adversely impact study participation or safety, conduct of the study, or interfere with pain assessments;
11. Active skin conditions such as dermatitis, allergy, eczema, psoriasis, or abnormal skin healing in any body area;
12. Patients who have tattoos, scars, or moles that in the opinion of the Investigator are likely to interfere with dosing or study assessments at any of the potential injection sites;
13. Depression of moderate severity or more on the Patient Health Questionnaire (PHQ-9 greater than or equal to 10) at the Screening visit;
14. History of psychotic symptoms requiring antipsychotic treatment, or history of a suicide attempt/s within 180 days prior to Screening;
15. Arterial or venous thrombus, myocardial infarction, hospital admission for unstable angina, treatment with cardiac angioplasty, or cardiac vessel stenting within 90 days prior to Screening;
16. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome-related illness, acute or history of chronic hepatitis B or C. Positive tests for HIV-1 or -2 antibodies, hepatitis B surface antigen, or hepatitis C antibodies;
17. Current medical or arthritic condition/s that could interfere with evaluation of the index joint including fibromyalgia, rheumatoid arthritis, or other inflammatory arthropathies;
18. Patient who has undergone arthroscopic or open surgery to the index joint/s within 180 days of Screening visit;
19. Patient who has undergone replacement surgery of the index joint/s within 180 days of Screening visit;
20. The placement of surgical hardware or other foreign body in the treatment joint/s within 180 days of Screening visit;
21. Use or intend to use any medications/products known to alter the absorption, metabolism, or elimination processes of the study drug, including but not limited to St. John's Wort, within 30 days prior to Screening visit, unless deemed acceptable by the Investigator (or designee);
22. Use or intend to use any prescription medications/products within 14 days prior to Screening, unless deemed acceptable by the Investigator (or designee). Note: hormone replacement therapy or oral, implantable, injectable, or intrauterine contraceptive concomitant medications are acceptable;
23. Use or intend to use slow-release medications/products considered to still be active within 14 days prior to Screening, unless deemed acceptable by the Investigator (or designee);
24. Use or intend to use any non-prescription medications/products including phytotherapeutic/herbal/plant-derived preparations within 14 days prior to Screening visit, unless deemed acceptable by the Investigator (or designee) and Sponsor, or assignee, has given their prior consent;
25. Patients who are unable or unwilling to cease the use of tobacco- or nicotine-containing products during the study duration and have used tobacco- or nicotine-containing products within 90 days prior to Screening visit;
26. Receipt of blood products within 60 days prior to Screening visit;
27. Donation of blood from 90 days prior to Screening, plasma from 14 days prior to Screening, or platelets from 42 days prior to Screening;
28. Poor peripheral venous access;
29. Are sponsor employees;
30. Have participated in a clinical study involving administration of an investigational drug in the past 90 days or 5 half-lives of the study drug, whichever is longer, prior to Screening visit;
31. Have participated in any trial of a device, supplement, cognitive/behavioural therapy, physiotherapy or active exercise study within 30 days prior to the Screening visit;
32. Have previously completed or withdrawn from this study or any other study investigating OLP-1002 or have previously received the study drug;
33. Patients who, in the opinion of the Investigator (or designee), should not participate in this study.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment- Emergent Adverse Events(Safety and Tolerability) of OLP-1002 in patients who have pain in a hip and/or knee joint | Monitored from Screening Visit till the end of the study visit(day 45).
  Number of participants with treatment-related adverse events as assessed by CTCAE
Safety and tolerability (Incidence of Treatment-Emergent Adverse Events) measure through Vital Sign- heart rate | Monitored from Screening Visit till the end of the study visit(day 45).
  Measured by result of the Vital Sign- heart rate
Safety and tolerability (Incidence of Treatment-Emergent Adverse Events) measure through Vital Sign- blood pressure | Monitored from Screening Visit till the end of the study visit(day 45).
  Measured by result of the Vital Sign- blood pressure
Safety and tolerability (Incidence of Treatment-Emergent Adverse Events) measure through Vital Sign- oral temperature | Monitored from Screening Visit till the end of the study visit(day 45).
  Measured by result of the Vital Sign- oral temperature
Safety and tolerability(Incidence of Treatment-Emergent Adverse Events) measure through 12-lead ECG | Monitored from Screening Visit till the end of the study visit(day 45).
  Measured by result of the ECG measurements and findings Parameters: QRS, ST segment, and QTcF.
Safety and tolerability(Incidence of Treatment-Emergent Adverse Events) measure through Physical exam | Monitored from Screening Visit till the end of the study visit(day 45).
  Measured by result of the physical exam which includes general appearance, head, ears, eyes, nose, throat, dentition, thyroid, chest (heart, lungs), abdomen, skin, neurological, extremities, back, neck, musculoskeletal, and lymph nodes.
Safety and tolerability(Incidence of Treatment-Emergent Adverse Events) measure through Clinical laboratory results | Monitored from Screening Visit till the end of the study visit(day 45).
  Measured by clinically significant change from baseline clinical laboratory results

SECONDARY OUTCOMES:
To evaluate the preliminary efficacy of OLP-1002 on pain, during the treatment and follow-up periods through WOMAC. The minimum and maximum values, and whether higher scores mean a better or worse outcome. | Monitored on Day 4, 8, 11, 15, 18, 25, 32 and 45.
  Measured by Western Ontario and McMaster Osteoarthritis Index (WOMAC) Pain, Stiffness and Physical Function Subscales together with Total WOMAC Score
To evaluate the preliminary efficacy of OLP-1002 on pain, during the treatment and follow-up periods through VAS. The minimum and maximum values, and whether higher scores mean a better or worse outcome. | Monitored on Day 4, 8, 11, 15, 18, 25, 32 and 45.
  Measured by Visual Analogue Scale (VAS)- Worst daily pain intensity
To characterize the pharmacokinetic (PK) profile of OLP-1002 trough concentration (Ctrough) | PK samples will be collected pre-dose on days Day 1, 8 and 15 as well as on Day 45
  Parameter: trough concentration (Ctrough); sample type used for these analysis: serum sample
To monitor the effects of multiple SC doses of OLP-1002 on Quality of Life (QoL) through Score (KOOS). The minimum and maximum values, and whether higher scores mean a better or worse outcome. | Monitored on Day 8, 15, 25, 32 and 45
  Measured by Change from Baseline in the Knee Injury and Osteoarthritis Outcome Score (KOOS)
To monitor the effects of multiple SC doses of OLP-1002 on Quality of Life (QoL) through Score (HOOS) QoL Subscale. The minimum and maximum values, and whether higher scores mean a better or worse outcome. | Monitored on Day 8, 15, 25, 32 and 45
  Measured by Change from Baseline in Hip Injury and Osteoarthritis Outcome Score (HOOS) QoL Subscale

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Ostor, Principal Investigator — Emeritus Research
Locations (4):
- Australia (4):
  - Paratus Clinical Research- Canberra Trial Clinic, Canberra, Australian Capital Territory
  - Paratus Clinical Research Western Sydney, Blacktown, New South Wales
  - Novatrials (Pendlebury Research), Newcastle, New South Wales
  - Emeritus Research, Camberwell, Victoria